CLINICAL TRIAL: NCT05149183
Title: Effect of Cervical Stability Training on Somatosensory Evoked Potential and Cervical Spine in Forward Head Posture
Acronym: FHP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003459
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Forward Head Posture
Keywords: cervical stability; somatosensory evoked potential; forward head posture

STUDY DESIGN:
Intervention Model Description: this trial has two groups, one experimental and one control
Who Masked: Participant, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical stability training (Experimental): cervical stability training will be received three times a week for eight weeks
  Interventions: Other: cervical stability training; Other: traditional treatment
- traditional treatment (Active Comparator): traditional treatment will be received three times a week for eight weeks
  Interventions: Other: traditional treatment

INTERVENTIONS:
Other: cervical stability training — cervical stability training will be contain three phases, each phase has six positions ( supine, forearms, sidelying, four point kneeling, sitting and standing position)
  Arms: cervical stability training
Other: traditional treatment — TENS, hot packs, stretching exercise of superficial neck muscles, and postural advice.

SUMMARY:
to investigate the effect of cervical stability training on somatosensory evoked potential and cervical spine in forward head posture

DETAILED DESCRIPTION:
The use of electronic tools is increasing in worldwide varieties and the attractiveness of these tools lead to variety of groups of people, especially teenagers, using them for prolonged period of time leading to increased musculoskeletal problems. Excessive use of smartphones for long period of time can lead to decreased postural control and forward head postur (FHP) as phone users maintain an abnormal alignment of the head and neck. The habit of repetitive use of computers, TV, mobile phones, and video games and even back packs forces the body to exhibit bad posture. The overall prevalence of FHP was reported to be 66% in computer based workers.

cervical stability training play a major role in treatment of forward head posture so this study will be conducted to investigate its role on craniovertebral angle, cervical range of motion, pain intensity level, functional disability, neck flexor and extensor muscles endurance, lordotic cervical curvature, somatosensory evoked potential in forward head patient.

ELIGIBILITY:
Inclusion Criteria:

Adult participant (18-to-40years old) with forward head posture, BMI 20-to-25 kg/m², The area of mechanical neck pain will defined to the cervical region, possibly with referred pain into the occipit, nuchal muscles, and shoulders, All patients will have chronic neck pain for more than 3 months, Craniovertebral angle of ˂ 49.

Exclusion Criteria:

Signs of serious pathology (e.g., rheumatoid diseases, ankylosing spondylitis), History of cervical spine surgery, History of trauma or fractures in cervical spine, Signs of cervical radiculopathy or myelopathy, Vascular syndrome such as vertebrobasilar insufficiency.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
somatosensory evoked potential | up to eight weeks
  somatosensory evoked potential will be measured by electromyograph device
craniovertebral angle | up to eight weeks
  craniovertebral angle will be measured photographically by surgimap program

SECONDARY OUTCOMES:
pain intensity level | up to eight weeks
  pain will be measured by visual analogue scale
functional disability | up to eight weeks
  disability will be measured by arabic neck disability index
cervical range of motion | up to eight weeks
  Phone application (clinometer) will used to measure cervical range of motion using smartphone (Infinix Note 5)
endurance test | up to eight weeks
  flexion and extension endurance will be measured using pressure biofeedback unit
cervical curvature | up to eight weeks
  digital x ray will be used to measure cervical curvature

CONTACTS AND LOCATIONS:
Locations (1):
- Salah Eid Ahmed Ali, Giza, Egypt